CLINICAL TRIAL: NCT06836999
Title: Using Deep Sedation vs. Conscious Sedation in Catheter Ablation in Patients With Atrial Fibrillation: Intraprocedural Management and Outcome Evaluation
Brief Title: Deep Sedation in Catheter Ablation of Atrial Fibrillation
Acronym: PRIORI-AF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Dalian Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TEMP-000758; ChiCTR2500096790 (Other: Chinese clinical trial registry)
Record Dates: First submitted 2025-02-16; First posted 2025-02-20 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2024-12

CONDITIONS: Atrial Fibrillation; Atrial Fibrillation, Paroxysmal or Persistent; Deep Sedations; Conscious Sedation
Keywords: deep sedation; conscious sedation; catheter ablation; atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Deep Sedation; Conscious Sedation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The present trial utilized a centralized randomization system (IWRS) to facilitate the competitive enrollment of study participants and treatment randomization grouping. The investigator (anesthesiologist) carries out the given treatment according to the grouping information of the study participants. Throughout the course of the study, the treatment groups were kept blind to the researchers, with the exception of the anesthesiologist, the sponsor, and the study participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DS group (Experimental): The CA procedure will be performed under deep sedation in the study group mainly with propofol for sedation and fentanyl for analgesic
  Interventions: Procedure: deep sedation
- CS group (Sham Comparator): The CA procedure will be performed under conscious sedation in the control group mainly with fentanyl.
  Interventions: Procedure: Conscious sedation

INTERVENTIONS:
Procedure: deep sedation — The deep sedation was inducted using atropine 0.5 mg iv administered 15 min before the procedure to avoid aspiration. In the EP lab, anesthesia preparation is performed, including invasive arterial blood pressure monitoring via puncture of the radial artery or brachial artery. Noninvasive BP monitoring every 5 minutes is also permitted. Subsequently, midazolam 1-2mg or accompanied with propofol 0.3-0.5 mg/kg is administered intravenously at the start of the CA procedure (i.e., femoral vein puncture), and fentanyl 25 µg is administered intravenously. Then, continuous titrated infusion of propofol 0.2-0.5mg/kg/h for anesthesia maintenance throughout the CA procedure. An additional iv fentanyl (25-50 µg) is administrated at the beginning of RF applications. Further boluses or additional drugs are administrated as needed to maintain analgesia during the procedure. The anesthesiologist is responsible for administering anesthesia and administering medication.
  Arms: DS group
Procedure: Conscious sedation — This protocol is aimed at analgesia, with local infiltration of lidocaine for femoral vein puncture followed by intravenous administration of fentanyl (1-2 ug/kg/h). The operator determines the dose of fentanyl and midazolam. A midazolam 1-5 mg bolus is administrated before electrical cardioversion is performed or when the patient is nervous.
  Arms: CS group

SUMMARY:
The current practice of anesthesia for atrial fibrillation catheter ablation （CA） procedure is inconsistent, including general anesthesia, deep sedation, and conscious sedation.Due to the nature of deep sedation, it has been continuously gaining its position as one of the crucial components in standard practices of atrial fibrillation ablation during the last decade. Currently, a considerable number of procedures have been done using conscious sedation. Previous studies explored the benefits obtained from the employment of deep sedation in AF ablation procedures, mainly focused on pain reduction and intra-procedural safety. However, the benefits on long-term rhythmic outcomes, peri-procedural safety as well as benefits on procedural parameters and peri-procedural experiences from patients/ablators/lab staff have yet not to be thoroughly studied. We plan to conduct a prospective, multicenter, randomized, controlled trial to evaluate the benefits of deep sedation in catheter ablation of paroxysmal and persistent AF in multiple prospective, i.e., quantified intraprocedural patients / physicians / lab staffs / mapper clinical specialist experiences, and the procedure safety.

ELIGIBILITY:
Inclusion Criteria:

● Patients diagnosed with AF (paroxysmal, persistent, or long-standing) at 18-75 years old who are eligible for the CA procedure

Exclusion Criteria:

* has received CA procedure for AF or atrial septal defect repair before enrollment
* left atrial diameter (LAD) ≥55 mm or thrombosis in the left atrium;
* eGFR<30mL/min/1.73㎡
* a history of cerebrovascular disease within the last three months (including stroke and transient ischemic attack [TIA])
* acute or severe systemic infection
* intolerant to sedation or with a history suggestive of sleep apnea
* BMI > 35 kg/㎡
* has contraindications to procedural sedation or refused to participate in this trial
* Congenital heart disease, thyroid dysfunction, severe hepatic insufficiency (Child-Pugh classification B-C), severe coagulation dysfunction (international normalized ratio (INR) > 1.5 or partial activated prothrombin time (APTT) prolonged by ≥ 10 seconds, or plasma prothrombin time (PT) prolonged by ≥ 3 seconds, or fibrinogen (Fib) ≤ 1.5 g/L), or active bleeding
* pregnant women, breastfeeding women or women who plan to become pregnant during the study period, those who have a positive pregnancy test result during the screening period
* life expectancy < 12 months
* those who have participated in other clinical drug trials within 3 months prior to enrollment
* those who are known to be allergic to any of the ingredients such as lidocaine, propofol, soybeans, peanuts, etc.
* those who, in the judgment of the investigator, are not suitable for this clinical study (e.g., not in line with the treatment that the research participants the treatment, research participant compliance, etc.).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1334 (Estimated)
Dates: Start 2025-03-03 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Rhythm outcomes | 4-12month post-ablation
  The primary effectiveness endpoint is the freedom from documented atrial arrhythmia (AF/AFL/AT lasting for over 30 seconds) recurrence monitored by ECG, 7-day ambulatory ECG, or equivalent cardiac monitoring from 4th to 12th month (9 months) after the procedure without taking I/III AADs. Patients who had to redo ablation or failed to discontinue I/III AADs after the blanking period are considered as primary endpoint

SECONDARY OUTCOMES:
Score of patients' intraprocedural experiences | during the CA procedure
  Questionnaires for patient：QoR-40 and Likelihood to recommend (LTR).
Score of ablators', staffs',nurse's intraprocedural experiences | during the CA procedure
  Likelihood to recommend (LTR) Questionnaire
respiratory system safety outcome | From the start of sedation to the end of the procedure
  the incidence of intraprocedural severe decrease in blood oxygenation (decrease in fingertip oxygen saturation to less than 90% or a >10% decrease in fingertip oxygen saturation from baseline)，apnea, respiratory depression, need for ventilator-assisted ventilation, and need for respiratory stimulant therapy
Rate of re-ablation acceptances | 4-12month post-ablation
  Rate of re-ablation acceptances if AF/AT recurrences.
Procedure time | during the CA procedure
  Procedure time (skin to skin), fluoroscopy, ablation time, etc.
The dosage of painkillers | during the CA procedure
  The dosage of painkillers
the incidence of regurgitation and aspiration and oral mucosal damage caused by oropharyngeal airway | From the start of sedation to the end of the procedure
  the incidence of regurgitation and aspiration and oral mucosal damage caused by oropharyngeal airway

CONTACTS AND LOCATIONS:
Overall Officials: Yunlong Xia, Ph.D, Principal Investigator — The First Affiliated Hospital of Dalian Medical University
Locations (16):
- China (16):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - NanFang Hospital, Guangzhou, Guangdong
  - Jiangsu Provincial Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - Qingdao Municipal Hospital, Qingdao, Shandong
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - Shanxi Cardiovascular Hospital, Taiyuan, Shanxi
  - Tianjin Chest Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - The Second Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang
  - Sir Rung Rung Shaw Hospital, Zhejiang University School Of Medicine, Hangzhou, Zhejiang
  - The Affiliated Hospital Of Medical School Of Ningbo University, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: No
To protect the privacy of subjects, the study data can be accessed by requesting from the PI.

REFERENCES:
- [Background] Grimaldi M, Quadrini F, Caporusso N, Troisi F, Vitulano N, Delmonte V, Di Monaco A. Deep sedation protocol during atrial fibrillation ablation using a novel variable-loop biphasic pulsed field ablation catheter. Europace. 2023 Aug 2;25(9):euad222. doi: 10.1093/europace/euad222. PMID 37470452
- [Background] Benzoni T, Agarwal A, Cascella M. Procedural Sedation. 2025 Mar 22. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK551685/ PMID 31869149